CLINICAL TRIAL: NCT07139197
Title: The Effect of a Cognitive Behavioral Approach-Based Psychoeducation Program on Cognitive Flexibility and Rumination in Elderly Individuals Living in Nursing Homes
Brief Title: The Effect of Cognitive Behavioral Therapy (CBT)-Based Psychoeducation on Cognitive Flexibility and Rumination in the Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Leyla ALTUN, Research Assistant, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AU-SBF-LA-01
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Cognitive Flexibility; Rumination; Elderly (People Aged 65 or More); Psychoeducation
Keywords: elderly; psychoeducation; cognitive flexibility; rumination; cognitive behavioral therapy
MeSH Terms: conditions — Rumination Syndrome

STUDY DESIGN:
Intervention Model Description: This study is planned to be conducted using a randomized controlled, pre-test-post-test, control group, and 1-month follow-up test experimental study design.To prevent contamination between groups, data collection for the intervention and control groups will be conducted at different times, except for the pre-test stage, which will be administered simultaneously by an independent assessor. The control group will not be subject to any intervention during the study period, but will be offered the psychoeducation programme after the study is completed if they wish.
Who Masked: Participant, Outcomes Assessor
Masking Description: During the pre-test phase, both the participants and the independent evaluators will be unaware of the group distribution. The allocation of group assignments will be determined subsequent to the completion of baseline assessments. Following randomisation, participants will be informed of the group distribution due to the nature of the psychoeducational intervention; however, the baseline assessment results will be conducted blindly.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group: Cognitive Behavioral Therapy (CBT)-Based Psychoeducation Program (Experimental): Participants in this group will receive a cognitive-behavioral psychoeducation program aimed at improving cognitive flexibility and reducing rumination. Pre-test assessments will be conducted before group allocation.
  Interventions: Behavioral: Cognitive Behavioral Approach-Based Psychoeducation Program
- Control Group: Usual Care (Standard Nursing Home Care) (No Intervention): Participants in this group will not be subject to any intervention during the study period. Pre-test assessments will be conducted by an independent evaluator simultaneously with the intervention group. Upon completion of the study, control group participants will be offered the opportunity to participate in the psycho-education program if they wish.

INTERVENTIONS:
Behavioral: Cognitive Behavioral Approach-Based Psychoeducation Program — Intervention Group: Cognitive Behavioral Approach-Based Psychoeducation Program Participants will receive a cognitive-behavioral psychoeducation program designed to improve cognitive flexibility and reduce rumination. The sessions include structured activities, discussions, and exercises based on cognitive-behavioral principles. Pre-test assessments will be conducted before group allocation.
  Control Group: No intervention will be provided during the study period. Participants will complete pre-test assessments administered by an independent evaluator. After the study concludes, control group participants will be offered the opportunity to participate in the psychoeducation program if they wish.
  Arms: Intervention Group: Cognitive Behavioral Therapy (CBT)-Based Psychoeducation Program

SUMMARY:
This study aimed to investigate the effect of psychoeducation on rumination and cognitive flexibility in elderly individuals residing in nursing homes. Cognitive Behavioral Therapy (CBT)-based psychoeducation has recently been applied to multiple specific groups around the world and in our country. In general, executive functioning skills and, more specifically, cognitive flexibility appear to be important for the ability to use certain CBT techniques; however, considering that these skills naturally decline with age, further research is needed. It is anticipated that the results of this study will contribute to applications in the field of psychiatric nursing.

DETAILED DESCRIPTION:
Aging causes neuroanatomical and physiological changes that affect cognitive processes such as memory, attention, and executive functions. Positive developments in healthcare worldwide, along with increasing socioeconomic levels and declining birth rates, have led to an increase in the elderly population. Our country, like many other countries around the world, is one of the rapidly aging countries. With the increase in the elderly population, the needs specific to the elderly are increasing, and it is inevitable to encounter a series of problems.

As age increases, the cognitive abilities of older adults decline. Research shows that working memory and long-term memory abilities decline, as do reasoning ability, processing speed, executive function, and attention control. As a result, individuals' quality of life, independence, and daily activities such as planning medication and grocery shopping may be negatively affected.

Cognitive flexibility plays a fundamental role in the ability to adapt to constantly changing environments and is associated with various goal-directed behaviors, including creativity, problem solving, multitasking, and decision making. Cognitive flexibility and the underlying processes (executive functions) have also been linked to self- and emotional regulation, as well as mental health outcomes. Cognitive flexibility refers to the ability to change one's cognitive organization, thinking, or attention in order to perceive, process, or respond to situations in different ways. The skills required for cognitive restructuring closely align with those related to cognitive flexibility. Cognitive flexibility encompasses the ability to generate diverse ideas, evaluate response alternatives, and modify behavior and cognition in response to changing environmental demands. These processes appear to be important for the successful implementation of cognitive restructuring, which requires the individual to identify negative automatic thoughts, generate evidence that contradicts these thoughts, and then produce a more adaptive or helpful way of interpreting the situation.

Rumination is associated with inflexible cognitive and emotional processes. Various characteristics of rumination-related thinking, including its negative value content, abstract level of interpretation, and passive approach to problem-solving, may also contribute to its maladaptive outcomes.

In order to successfully carry out daily activities, it is necessary to be able to flexibly switch from one behavior to another. This skill is referred to as cognitive flexibility. Individuals who ruminate experience cognitive rigidity by getting stuck on a certain thought and find it difficult to change the behaviors they focus on. At the same time, cognitive rigidity is also thought to be the underlying cause of repetitive thinking patterns in rumination. It is well known that mental rumination, a negative and evaluative mode of repetitive thinking, is the main psychological process that accelerates and sustains depressive mood. In this context, rumination may be a variable that predicts cognitive flexibility. In particular, perseverative thinking styles have been found to negatively affect the ability to learn cognitive restructuring. Further research is needed to clarify whether older adults with weak cognitive flexibility can develop their cognitive restructuring skills through repetition rather than treatment, or whether alternative skills should be considered.

To date, there has been little research examining whether declines in cognitive abilities have an impact on overall treatment outcomes or the acquisition of specific therapeutic skills. Given the aging of the world's population, it is important to focus more research on understanding the impact of age-related cognitive changes in older adults on the treatment of mental health problems. This study will focus on cognitive flexibility and rumination, which are processes responsible for producing changes in behavior and thought in dynamic contexts and are subject to fluctuations and rapid changes.

ELIGIBILITY:
Inclusion Criteria:

* Be 65 years of age or older,
* Be willing to participate in the study,
* Not have hearing or vision problems that would prevent understanding the training to be provided,
* Have communication and comprehension skills,
* Be literate,
* Have a Standardized Mini Mental Test score between 25 and 30 points.

Exclusion Criteria:

* Having any hearing or vision problems.
* Having physical, neurological, or psychological health problems that could disrupt group harmony and integrity.
* Having an illness or problem that could prevent them from responding to the measurement tools used in the study.
* Having a Standardized Mini Mental Test score below 25.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-09-15 (Estimated); Study Completion 2026-06-15 (Estimated)

PRIMARY OUTCOMES:
Cognitive Flexibility Inventory | 8 weeks
  The inventory was adapted into Turkish. The five-point Likert-type inventory consists of two subscales, "alternatives" and "control," and 20 items. The "alternatives" subscale consists of statements regarding the possibility of finding alternative solutions to difficult situations or alternative explanations for life circumstances and human behavior. The "control" subscale consists of statements about the controllability of difficult situations. The lowest possible score on the inventory is 20, and the highest possible score is 100. Items 2, 4, 7, 9, 11, and 17 of the scale are reverse-coded. High scores on the inventory indicate high cognitive flexibility. In the Turkish version of the inventory, the Cronbach's alfa coefficient (Cronbach's alpha) was calculated as .90 for the entire inventory, .90 for the alternatives subscale, and .84 for the control subscale.
Self-Critical Rumination Scale | 8 weeks
  The scale was adapted into Turkish. The scale is a unidimensional scale with a 4-point Likert scale (1 = Never, 2 = Somewhat, 3 = Mostly, 4 = Completely). The scale's fit indices were found to be chi-square/degrees of freedom (x²/df) = 3, Root Mean Square Error of Approximation (RMSEA) = .08, Tucker-Lewis Index (TLI) = .93, Comparative Fit Index (CFI) = .94, and Standardized Root Mean Square Residual (SRMR) = .04. In criterion-related validity, the correlation between the Ruminative Responses Scale short form (RRS) and the RRS was found to be r = .73, with the obsessive thinking subscale r = .73 and the deep thinking subscale r = .68. The internal consistency coefficient of the scale was Cronbach's alfa coefficient (Cronbach's alpha) = .89, and the test-retest reliability coefficient, measured five weeks apart, was .83.

SECONDARY OUTCOMES:
Standardized Mini Mental Test (SMMT) | 1 weeks
  A standardized version of the test was created, taking into account sociocultural differences in our country. This test consists of five subcategories-orientation, memory, attention and calculation, recall, and language-and 11 items. It is scored out of a total of 30 points, with each correct answer earning one point. The lowest possible score is 0, and the highest possible score is 30. A score between 0 and 12 indicates severe cognitive impairment, a score between 13 and 22 indicates moderate cognitive impairment, a score between 23 and 24 indicates early-stage cognitive impairment, and a score between 25 and 30 indicates no cognitive impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Kars Huzurevi Yaşlı Bakım ve Rehabilitasyon Merkezi / Kars Huzur Evi Elderly Care and Rehabilitation Center, Kars, Center, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No